CLINICAL TRIAL: NCT03445819
Title: A Prospective Randomized Trial of Non-operative Versus Operative Management of Patella Fractures in the Elderly
Brief Title: Patella Fracture : A Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Patella RCT 2018
Record Dates: First submitted 2018-02-13; First posted 2018-02-26 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Patella Fracture; Aging
Keywords: Patella Fracture, elderly
MeSH Terms: conditions — Patella Fracture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Data analysts will be blinded to the study treatment.Wherever possible, outcome assessors will be blinded to the study treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Surgical Treatment (Other): Open reduction and internal fixation (ORIF) of the patellar fracture will be performed using screws, wires, pins, or plate fixation at the discretion of the treating surgeon. The trial is designed in a pragmatic fashion to allow participating surgeons from the multiple participating sites to perform fixation as per the standard of care at their institution. Post-operative care will include standard-of-care antibiotics and deep vein thrombosis (DVT) prophylaxis, both prescribed at the discretion of the attending surgeon.
  Interventions: Procedure: Group A: Surgical Treatment
- Group B: Conservative Treatment (Other): Patients randomized to non-operative treatment will receive identical treatment to the operative group, minus the surgery. Patients will be weight bearing as tolerated immediately in a removable knee immobilizer, with progressive range-of-motion exercises begun at two weeks following randomization
  Interventions: Other: Group B: Conservative Treatment

INTERVENTIONS:
Procedure: Group A: Surgical Treatment — Open reduction and internal fixation (ORIF) of the patellar fracture will be performed using screws, wires, pins, or plate fixation at the discretion of the treating surgeon
  Arms: Group A: Surgical Treatment
Other: Group B: Conservative Treatment — Patients randomized to non-operative treatment will receive identical treatment to the operative group, minus the surgery.
  Arms: Group B: Conservative Treatment

SUMMARY:
This is a multi-centre, randomized controlled trial comparing operative and non operative treatment for displaced patella fractures in elderly, low-demand patients.

DETAILED DESCRIPTION:
Patients with a displaced patellar fracture who meet the inclusion criteria and provide consent will be randomized to one of the two treatment arms. One group (Group A) will receive standardized non-operative treatment with immediate weight-bearing as tolerated in a knee immobilizer and early ROM exercises begun at 2 weeks post injury. The other group (Group B) will receive ORIF of their displaced patellar fracture with a standardized post-operative protocol.

Post-operative rehabilitation will be standardized across both groups. Patients will be weight bearing as tolerated immediately in a removable knee immobilizer, with progressive range-of-motion exercises begun at two weeks following surgery or randomization. The knee immobilizer will be used full-time (with the exception of removal for physiotherapy and bathing) for 6 weeks after surgery or randomization. At six weeks post-treatment, patients will be allowed to perform active extension and will initiate progressive strengthening exercises of the extensor mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 65 years of age or older and ambulatory prior to injury (with or without walking aids).
* Closed fracture of the patella displaced by 5 mm or greater (Displacement will be determined by measuring the widest displacement on any x-ray view with the knee in full extension).
* The patient scores between 3 and 6 on the Clinical Frailty Scale. This score corresponds to a low-demand patient who is ambulatory and functionally independent
* Within 14 days of injury, the patient is able to perform a straight leg raise with less than 30 degrees of extensor lag.
* Able to read and understand the study consent form document.
* Willing and able to sign consent, follow the study protocol and attend follow-up visits.

Exclusion Criteria:

* Associated extremity injuries or polytrauma injuries that would otherwise require surgery or interfere substantially with rehabilitation or outcome in the opinion of the investigator.
* Neurovascular injuries at the level of the knee requiring surgery.
* Pathologic fractures.
* Periprosthetic fractures, or other knee surgery which would contra-indicate inclusion in the study (e.g. previous patella ORIF or previous surgery involving patella such as patella tendon or quads repair).
* Medical contra-indication to surgery.
* Likely problems, in the judgment of the investigators, with maintaining follow-up (e.g. patients with no fixed address, intellectually challenged patients without adequate support, etc.).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee injury and Osteoarthritis Outcome Score (KOOS) | 1 year after injury
  A self-administered questionnaire that assesses five outcomes: pain, symptoms, activities of daily living, sport and recreation function, and knee-related quality of life. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.

SECONDARY OUTCOMES:
Visual Analogue Pain Scale (VAS) | 1 year after injury
  VAS consists of a straight line with the endpoints defining extreme limits of pain, ranging from 'no pain at all' (zero) to 'pain as bad as it could be' (10)
Range of Motion | up to 24 months
  Measurement of flexion and extension

OTHER OUTCOMES:
TUG Test | up to 24 months
  Timed Up and Go test

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Nauth, MD, FRCS (C), Principal Investigator — Unity Health Toronto; Jeremy Hall, MD, FRCS(C), Principal Investigator — Unity Health Toronto
Locations (3):
- Canada (3):
  - London Health Sciences Centre, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
No plan

REFERENCES:
- [Derived] Sayum Filho J, Lenza M, Tamaoki MJ, Matsunaga FT, Belloti JC. Interventions for treating fractures of the patella in adults. Cochrane Database Syst Rev. 2021 Feb 24;2(2):CD009651. doi: 10.1002/14651858.CD009651.pub3. PMID 33625743